CLINICAL TRIAL: NCT03405194
Title: An Open-Label, Randomized Comparison of Elvitegravir-Cobicistat-Tenofovir Alafenamide-Emtricitabine Versus Efavirenz-Tenofovir Disoproxil Fumarate-Lamivudine in Patients Starting Antiretroviral Therapy on the Day of HIV Diagnosis
Brief Title: Same-Day Treatment With Genvoya vs. EFV/TDF/3TC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Haiti gained access to dolutegravir as first-line ART, so we cancelled the study before any patient was enrolled (we didn't want SOC group to receive EFV)
Sponsor: Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic (Other)
Collaborators: Gilead Sciences (Industry); Brigham and Women's Hospital (Other); Weill Medical College of Cornell University (Other); Analysis Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IN-US-292-4500
Record Dates: First submitted 2017-12-24; First posted 2018-01-23 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Same-Day ART; Genvoya; Efavirenz
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — elvitegravir; Cobicistat; Racivir; efavirenz

STUDY DESIGN:
Intervention Model Description: Same-Day ART with Genvoya vs. EFV/TDF/3TC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Elvitegravir-Cobicistat-TAF-FTC (Experimental): Elvitegravir 150mg po QD Cobicistat 150 mg po QD TAF 10 mg po QD FTC 200 mg QD
  Interventions: Drug: Elvitegravir, Cobicistat, TAF, FTC
- EFV-TDF-3TC (Active Comparator): EFV 600 mg po QD TDF 300 mg po QD 3TC 300 mg po QD
  Interventions: Drug: Efavirenz, TDF, and 3TC

INTERVENTIONS:
Drug: Elvitegravir, Cobicistat, TAF, FTC — Started on day of HIV diagnosis
  Arms: Elvitegravir-Cobicistat-TAF-FTC
Drug: Efavirenz, TDF, and 3TC — Started on day of HIV diagnosis
  Arms: EFV-TDF-3TC

SUMMARY:
Randomized, open-label study comparing Elvitegravir-Cobicistat-Tenofovir Alafenamide-Emtricitabine (Genvoya) vs. Efavirenz-Tenofovir Disoproxil Fumarate-Lamivudine (EFV-TDF-3TC) in patients starting ART on the day of HIV diagnosis.

DETAILED DESCRIPTION:
Patients with WHO Stage 1 or 2 disease at HIV diagnosis will be randomized in a 1:1 ratio to either the Genvoya group or the EFV-TDF-3TC group. ART will be initiated on the day of HIV diagnosis. Participants who are found to have a contraindication to their assigned treatment regimen will change ART, and be classified as a failure for their assigned treatment arm. Participants in the EFV-TDF-3TC group with CrCl of 30-50 mL/minute, or with baseline mutations that significantly reduce the susceptibility of EFV will switch to Genvoya. Participants in the Genvoya group who are diagnosed with TB after enrollment will be switched to an ART regimen that can be administered with rifampin. If the study physician determines that a treatment change is indicated due to intolerability or side effects, the relevant clinical data will be presented to a safety committee that is blinded to group assignment. The ART regimen will be changed if the safety committee determines that it is indicated, and the participant will be considered a failure to their assigned treatment group. Patients will be followed for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of positive HIV status (test conducted at GHESKIO);
* At least 18 years of age;
* Unaware of HIV diagnosis prior to date of enrollment, and ART-naïve;
* Ability and willingness to give written informed consent;
* Ready to initiate same-day ART, according to two criteria: (1) HIV medication readiness questionnaire; and (2) social worker assessment;
* WHO Stage 1 or 2 disease, as defined by the following conditions: asymptomatic; persistent generalized lymphadenopathy; unexplained weight loss (under 10%); recurrent upper respiratory tract infections; herpes zoster; angular chelitis; recurrent oral ulcerations; papular pruritic eruptions; seborrheic dermatitis; or fungal nail infections.
* Female participants may be enrolled if they are either: (1) post-menopausal; (2) physically incapable of becoming pregnant due to tubal ligation, hysterectomy, or bilateral oophorectomy; or (3) are of childbearing potential, and agree to use one of the following methods to avoid pregnancy throughout the duration of the study:

Complete abstinence from intercourse; Double barrier method, such as male condom/spermicide, male condom/diaphragm, or diaphragm/spermicide; Hormonal contraception plus a barrier method; Intrauterine device (IUD); Male partner sterilization (if participant has only one sexual partner);

Exclusion Criteria:

* Pregnancy or breastfeeding at the screening visit;
* Active drug, alcohol use, or mental condition that would interfere with the ability to adhere to study requirements, in the opinion of the study physician;
* World Health Organization Stage 3 or 4 disease, as defined by the following conditions: unexplained severe weight loss (over 10% of presumed or measured body weight); unexplained chronic diarrhea for longer than 1 month; unexplained persistent fever (intermittent or constant for longer than 1 month); persistent oral candidiasis; oral hairy leukoplakia; pulmonary tuberculosis; severe bacterial infections (e.g. pneumonia, empyema, meningitis, pyomyositis, bone or joint infection, bacteremia, severe pelvic inflammatory disease); or acute necrotizing ulcerative stomatitis, gingivitis or periodontitis.
* Clinical evidence of cirrhosis (ascites or encephalopathy);
* Anticipated need for hepatitis C therapy during the study period;
* Baseline CrCl <30 mL/minute by the Cockcroft-Gault equation (late exclusion, as creatinine results will not be available at the time of enrollment);
* Either the K65R mutation or more than 3 thymidine analogue mutations on baseline resistance testing (late exclusions, after baseline resistance results are available).
* Planning to transfer care to another clinic during the study period;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
48-week viral suppression | 48 weeks after enrollment
  To compare the proportion of participants who are retained in care with a plasma HIV-1 RNA level <200 copies/ml

SECONDARY OUTCOMES:
12-week viral suppression | 12 weeks after enrollment
  Proportion of participants who are retained in care with a plasma HIV-1 RNA level <200 copies/ml
Baseline resistance to ART medications | Baseline
  Genotypic resistance to EFV and/or nucleoside reverse transcriptase inhibitors
Change in CD4 count | 48 weeks after enrollment
  Median change in CD4 count over the study period (baseline to 48 weeks)
Virologic failure | 48 weeks after enrollment
  Proportion of patients meeting the WHO definition for ART treatment failure over the study period
Adverse events | 48 weeks after HIV testing
  Proportion of participants with a new Division of AIDS Grade 3 or 4 adverse event or laboratory abnormality that is at least a one-grade increase from baseline
Neurologic or psychiatric adverse event | 48 weeks
  Proportion of participants with a new Division of AIDS Grade 1 to 4 neurologic or psychiatric disorder that is at least a one-grade increase from baseline
Sleep Quality | 4, 12, 24, and 48 weeks after enrollment
  Mean scores on the Pittsburgh Sleep Quality Index
Depression | 4, 12, 24, and 48 weeks after enrollment
  Mean scores on the Patient Health Questionnaires (PHQ-9) Questionnaire
Change in ART drugs | 48 weeks after HIV testing after enrollment
  Proportion of participants who discontinue any drug in the original ART regimen

CONTACTS AND LOCATIONS:
Overall Officials: Jean W Pape, MD, Principal Investigator — Haitian Group for the Study of Kaposi's Sarcoma and Opportunistic; Serena P Koenig, MD, Principal Investigator — Brigham and Women's Hospital